CLINICAL TRIAL: NCT03493204
Title: Tackling 30-day Readmissions in Patients With Cirrhosis: The SALTYFOOD Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Elliot B. Tapper, Assistant Professor of Internal Medicine, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUM00141457
Record Dates: First submitted 2018-04-03; First posted 2018-04-10 (Actual); Last update posted 2019-08-30 (Actual); Status verified 2019-08

CONDITIONS: Hepatic Encephalopathy; Ascites; Liver Diseases; Cirrhosis
Keywords: Hepatic Encephalopathy; Ascites; Liver Diseases; Cirrhosis
MeSH Terms: conditions — Hepatic Encephalopathy; Ascites; Liver Diseases; Fibrosis | interventions — Nutrition Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Home-delivered, salt restricted (Experimental): Meal description: salt-restricted (1500 mg to 2000 mg daily), > 2100 kilocalorie, high protein (>80 g daily) in addition to receiving standard pamphlet receipt
  Interventions: Other: Meal delivery
- Dietary Advice (Active Comparator): Standard of care, advice on salt-restriction using standard pamphlet receipt
  Interventions: Other: Standard pamphlet with Dietary Advice

INTERVENTIONS:
Other: Meal delivery — The food will be pre-packaged for storage and patient will prepare these meals at home
  Arms: Home-delivered, salt restricted
Other: Standard pamphlet with Dietary Advice — Explains how to maintain a low-sodium diet
  Arms: Dietary Advice

SUMMARY:
The purpose of this study is to determine the feasibility of a home meal delivery program for patients with cirrhosis and ascites and to determine the effectiveness of a salt-restricted (2 gram sodium) meal delivery program in reducing the need for therapeutic paracenteses and/or all-cause re-admissions for these patients. Many patients with cirrhosis don't have enough nutrients in the body and are frail and these meals may help them maintain a good diet and lead to improved quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Adult 18 years or older of age
* Clinical diagnosis of cirrhosis with ascites. Diagnosis of cirrhosis will be based upon:

  1. liver biopsy, OR
  2. history of cirrhosis complication: ascites, variceal bleeding, hepatic encephalopathy, OR
  3. 2 of the following 4 criteria: i. Ultrasound (US), computerized axial tomography (CT) or Magnetic Resonance Imaging (MRI) imaging findings of cirrhosis (cirrhotic appearing liver, splenomegaly, varices, ascites) ii. Fibroscan liver stiffness score >13 kPa iii. Laboratory testing: Aspartate Aminotransferase (AST)/platelet ratio index (APRI) >2.0 iv. CT, MRI or Esophagogastroduodenoscopy (EGD) showing presence of esophageal varices
* 3) At least one of the following: Any cause hospitalization within 90 days OR outpatient therapeutic paracentesis within 30 days

Exclusion Criteria:

* Language barriers that cannot be surmounted with in-person interpreters
* Estimated life expectancy < 3 months
* Pregnancy (self-reported)
* Unable or unwilling to provide consent
* History of liver transplant
* Planned discharge to nursing facility
* Anuria or serum creatinine > 2.0 mg/dL
* Uncontrolled hepatic encephalopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2018-04-24 (Actual); Primary Completion 2019-08-19 (Actual); Study Completion 2019-08-19 (Actual)

PRIMARY OUTCOMES:
Number of therapeutic paracenteses | From date of randomization until 12 weeks
  Number of paracenteses

SECONDARY OUTCOMES:
Change in Quality of life | baseline, week 12
  Measured by Ascites Symptom Inventory (ASI-7). This is a 7 question scale that measures the subject's symptoms with a value from 0-4 (0=does not apply / 4=very strong applies). The higher the subject's score the worse the subject's symptoms. The mean change will be compared between groups.

OTHER OUTCOMES:
Number of hospital-bed days in 12 weeks | From date of randomization until 12 weeks
  The number of days the participants were hospitalized after randomization
Change in diuretic dose | baseline, week 12
  The dose amount changes the participant's medications that are considered diuretics
Change in frailty measures | baseline, week 12
  Change in the hand grip strength using a hand-held dynamometer. The device will be squeezed 3 times with their dominant hand and the force measured in kilograms. The best recorded value (highest force number) will be their value.
Change in frailty measures | baseline, week 12
  Change in time taken to walk 5 meters (walk speed measured in meters per second)
Quality of life | baseline, week 12
  Change in Visual Analog Scale. The subject selects how their health is today by marking an X on the scale from 0-100; 0= worst imaginable health state / 100= best imaginable health state

CONTACTS AND LOCATIONS:
Overall Officials: Elliot Tapper, Principal Investigator — University of Michigan
Locations (1):
- The University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Undecided